CLINICAL TRIAL: NCT02678091
Title: Contribution of the Quantitative Analysis of the Ultrasound Exam With Doppler for the Etiological Diagnosis of Orbital Masses (PUCE)
Brief Title: Ultrasound Exam With Doppler for the Etiological Diagnosis of Orbital Masses (PUCE)
Acronym: PUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALR_2015_40
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Tumor of the Orbit
MeSH Terms: conditions — Orbital Neoplasms | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Patients with an orbital mass
  Interventions: Device: Ultrasound exam with Doppler

INTERVENTIONS:
Device: Ultrasound exam with Doppler — Ultrasound exam of the orbit

SUMMARY:
Orbital masses develop at the expense of the orbital structures lacrimal glands, oculomotor muscles, optic nerve, meningeal spaces, peripheral nerves, bone wall, orbital fat, lymphoid structures or vascular structures. These masses can be tumors, benign or malignant, or pseudotumor, mainly represented by specific or non-specific orbital inflammation.

Pathology is of considerable importance for the diagnosis and the treatment of those masses. However, biopsy or surgical resection of the orbital masses is sometimes difficult and dangerous outside expert centers.

The identification of a non-invasive technique for distinguishing tumors from pseudotumors, thus avoid in some cases a biopsy, would be a major contribution for the patients.

Quantitative analysis of the ultrasound exam with doppler of those masses could identify diagnostic criteria, especially for the lacrimal gland, easily explorable.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 years or more
* with an orbital mass for which a biopsy and/or a surgical removal is planned
* before surgery or biopsy

Exclusion Criteria:

* pregnancy
* breast feeding
* patient under a legal protection procedure
* patient denying to participate to the study
* lack of affiliation to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity, expressed as a percentage, of the ultrasound exam with Doppler, the pathological exam being the gold standard | One month
Specificity, expressed as a percentage, of the ultrasound exam with Doppler, the pathological exam being the gold standard | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided